CLINICAL TRIAL: NCT01032369
Title: The Additive Effect of Cognitive Behavioral Treatment - CBT to Conventional Weight Loss Intervention Program for Young Adults With Intellectual Disabilities
Brief Title: The Additive Effect of Cognitive Behavioral Treatment (CBT) to Conventional Weight Loss Intervention Program for Young Adults With Intellectual Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TASMC-09-NV-587-CTIL
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Overweight; Obesity; Learning Disability
Keywords: Over-weight or obese subjects with learning disability who have completed "Nitzan Onim" two-year training program and live in housing within the community
MeSH Terms: conditions — Overweight; Obesity; Learning Disabilities | interventions — Exercise; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Experimental): with behavioral intervention-CBT.
  Interventions: Other: Nutritional intervention, physical activity and behavioral treatment
- Without CBT (Other): Without behavioral intervention-CBT
  Interventions: Other: Nutritional intervention and physical activity

INTERVENTIONS:
Other: Nutritional intervention and physical activity — Nutritional intervention:
  Subjects will be asked to attend weekly nutritional group's sessions and individual meetings with the dietician for nutritional treatment and follow up.
  Physical activity:
  All participants will be engaged in physical activity comprising 45-60 min training sessions 3 times a week (gym or walking).
  Arms: Without CBT
Other: Nutritional intervention, physical activity and behavioral treatment — Nutritional intervention:
  Subjects will be asked to attend weekly nutritional group's sessions and individual meetings with the dietician for nutritional treatment and follow up.
  Physical activity:
  All participants will be engaged in physical activity comprising 45-60 min training sessions 3 times a week (gym or walking).
  Behavioral treatment:
  This group will undergo behavioral treatment focusing on self control techniques using the CBT technique (cognitive behavioral therapy) which will be conducted by a clinical psychologist from "ONIM" in weekly group sessions.
  Arms: CBT

SUMMARY:
In this randomized case control study we will evaluate the additive effect of psychological intervention, i.e CBT-cognitive behavioral treatment in a multi-strategy weight loss program composed of physical activity intervention and nutritional programme.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with over-weight or obese subjects with learning disability who have completed "Nitzan Onim" two-year training program and live in housing within the community
* Subjects who sign an informed consent

Exclusion Criteria:

* Subjects with out over-weight or obese subjects with out learning disability subjects who have no completed "Nitzan Onim" two-year training program and live in housing within the community

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of behavioral intervention-CBT on weight loss program (nutrition counselling and physical activity). | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel